CLINICAL TRIAL: NCT00882648
Title: The Effect of Fetal Gender on Maternal Substance Abuse Treatment
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lauren M. Jansson, Associate Professr of Pediatrics Johns Hopkins University School of Medicine, National Institute on Drug Abuse (NIDA)
Other Study IDs: 19524; R01DA019934 (NIH)
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Drug Dependence; Pregnancy
Keywords: Drug dependence during pregnancy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Drug dependent women: All drug dependent women enrolled in comprehensive substance abuse treatment at the Center for Addiction and Pregnancy of Johns Hopkins University between 2004 and 2009; retrospective chart review.

SUMMARY:
Previous studies by this team of investigators has determined that male infants are more likely to display more severe neonatal abstinence syndrome (NAS) as a result of maternal opioid use during pregnancy (Jansson, 2007)and there is appears to be a gender-related biologic vulnerability to NAS expression (Jansson, 2009, submitted). The proposed study explores the relationship between fetal gender and substance abuse treatment outcomes among a population of women in comprehensive substance abuse treatment to explore the possibility of a psychosocial vulnerability among drug exposed male fetuses as opposed to female fetuses. Women in substance abuse treatment are a group at high risk for current exposure to violence, usually at the hands of significant others, and having a history of sexual abuse as a child, usually resulting from contact with a male family member. Therefore, they often have difficult relationships with men. At the Center for Addiction and Pregnancy (CAP), a 2006 study revealed that among a group of 715 pregnant women, reports of the exposure to violence was very high. Their rates of lifetime abuse ranged from 72.7% for physical abuse to 44.5% for sexual abuse. Rates of abuse remained high during their current pregnancy, ranging from 20% for physical abuse to 7.1% for sexual abuse (Velez, 2006). The abuse was very often at the hands of partners or other male family member perpetrators. We hypothesize that women carrying male fetuses will be less likely to remain complaint in drug treatment or abstinent from illicit drug use, while women carrying female fetuses may be more likely to remain drug abstinent and treatment compliant. If supported, this theory has the potential to inform fetal gender specific treatment for pregnant drug dependent women. Additionally, we seek to support the previously documented link between male gender and more severe expression of NAS, and explore the relationship between other maternal prescribed drug use (i.e. psychotropic medications) and severity of NAS expression.

ELIGIBILITY:
Inclusion Criteria:

* All CAP clients who either experience a pregnancy loss, or deliver an infant while in treatment at CAP between the years 7/1/03 and 6/30/08

Exclusion Criteria:

* All CAP clients who depart CAP treatment prior to pregnancy loss or birth during that time period

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women enrolled in comprehensive substance abuse treatment at the Center for Addiction and Pregnancy (CAP) between 2004 and 2009
Sampling Method: Non-Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Compliance with substance abuse treatment group and individual sessions and ability to maintain abstinence from illicit drug use | 1.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Addiction and Pregnancy, Baltimore, Maryland, United States